CLINICAL TRIAL: NCT02839850
Title: Multi-Center Clinical Evaluation of the ATTUNE Cementless Rotating Platform Total Knee Arthroplasty
Brief Title: 14022 ATTUNE Cementless RP Clinical Performance Evaluation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14022
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis
Keywords: Arthroplasty; replacement; Knee; function; radiographic; survivorship
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Masking Description: An independent radiographic reviewer will be assessing all radiographs from the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- ATTUNE Cementless RP TKA (Experimental): Subjects will receive a cementless, rotating platform total knee arthroplasty
  Interventions: Device: Cementless Total Knee Arthroplasty

INTERVENTIONS:
Device: Cementless Total Knee Arthroplasty — Patients will undergo a primary total knee replacement using one of the two configurations of the ATTUNE Cementless knee (CR RP or PS RP)

SUMMARY:
The primary objective of this study is to examine the change from pre-operative baseline to two year postoperative functional performance improvement for the ATTUNE primary, cementless TKA RP system as measured with the KOOS questionnaire (KOOS-ADL sub-score). This will be carried out for two configurations: cruciate retaining rotating platform (ATTUNE Cementless CR RP) and posterior stabilized rotating platform (ATTUNE Cementless PS RP).

DETAILED DESCRIPTION:
The secondary objectives of this study are:

* Evaluate change from preoperative baseline in post-operative outcomes using additional patient reported measures at 2 years: PKIP (overall and sub-scores), KOOS (overall and sub-scores), AKS and EQ-5D-3L.
* Evaluate change from preoperative baseline in pain and satisfaction over time as measured using a modified VAS Pain Score (discrete numbers rather than a continual scale) at 2yr.
* Evaluate type and frequency of Adverse Events
* Evaluate survivorship of the ATTUNE Primary Cementless TKA system for the CR RP and PS RP configurations using Kaplan-Meier survival analysis at 2yr and 5yrs.
* Evaluate primary, cementless ATTUNE TKA fixation through zonal radiographic analysis of the bone-implant interface at 6wk, 6mo, 1yr, and 2yr after surgery.
* Evaluate any changes in anatomic tibiofemoral, femoral component and tibial component alignment at 2 years compared to the first postoperative radiographs.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female and between the ages of 22 and 80 years at the time of surgery, inclusive.
* Subject was diagnosed with NIDJD.
* Subject, in the opinion of the Investigator, is a suitable candidate for cementless primary TKA using the devices described in this CIP with either resurfaced or non-resurfaced patellae.
* Subject that is willing to give voluntary, written informed consent to participate in this clinical investigation and authorize the transfer of his/her information to the Sponsor
* Subject is currently not bedridden
* Subject, in the opinion of the Investigator, is able to understand this clinical investigation and is willing and able to perform all study procedures and follow-up visits and co-operate with investigational procedures.
* Subject is able to read, and comprehend the Informed Consent Document as well as complete the required PROs in either English or one of the available translations.

Exclusion Criteria:

* The Subject is a woman who is pregnant or lactating.
* Contralateral knee has already been enrolled in this study .
* Subject had a contralateral amputation.
* Previous partial knee replacement (unicompartmental, bicompartmental or patellofemoral joint replacement), patellectomy, high tibial osteotomy or primary TKA in affected knee.
* Subject is currently diagnosed with radicular pain from the spine that radiates into the limb to receive TKA.
* Subject has participated in a clinical investigation with an investigational product (drug or device) in the last three (3) months.
* Subject is currently involved in any personal injury litigation, medical-legal or worker's compensation claims.
* Subject, in the opinion of the Investigator, is a drug or alcohol abuser (in the last 5 years) or has a psychological disorder that could affect their ability to complete patient reported questionnaires or be compliant with follow-up requirements.
* Subject was diagnosed and is taking prescription medications to treat a muscular disorder that limits mobility due to severe stiffness and pain such as fibromyalgia or polymyalgia.
* Subject has a significant neurological or musculoskeletal disorder(s) or disease that may adversely affect gait or weight bearing (e.g., muscular dystrophy, multiple sclerosis, Charcot disease).
* Subject is suffering from inflammatory arthritis (e.g., rheumatoid arthritis, juvenile rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus, etc.).
* Subject has a medical condition with less than five (5) years life expectancy.
* Uncontrolled gout

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Patient-reported Outcome: Knee Injury and Osteoarthritis Outcome Score Activities of Daily Living (KOOS ADL) | Minimum 2 years (670-1033 days after surgery)
  The Knee injury and Osteoarthritis Outcome Score (KOOS) is a patient self-administered questionnaire that consists of 42 questions and include the WOMAC Osteoarthritis index. The KOOS consists of 5 subscales: pain, other symptoms, activities of daily living (ADL), sport and recreational function and knee related quality of life. Each question has 5 Likert-like response options. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.

SECONDARY OUTCOMES:
Patient-reported Outcome: Pre-surgical/Post-surgical Patient's Knee Implant Performance (PKIP) | Minimum 2 years (670-1033 days after surgery)
  The Pre Surgical and/or Post-surgical Patient's Knee Implant Performance (PKIP) questionnaire is a patient self-administered questionnaire that consists of 25 questions relating to the patient's awareness of their knee. Questions include the patient's self-confidence about the current status of their knee performance, stability, and overall satisfaction. Each question has a 5, 6 or 10 Likert- like response option.
Patient-reported Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) | Minimum 2 years (670-1033 days after surgery)
  The Knee injury and Osteoarthritis Outcome Score (KOOS) is a patient self-administered questionnaire that consists of 42 questions and include the WOMAC Osteoarthritis index. The KOOS consists of 5 subscales: pain, other symptoms, activities of daily living (ADL), sport and recreational function and knee related quality of life. Each question has 5 Likert-like response options. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Combination of Patient-reported and Clinical-reported Outcome: Knee Society 2011 | Minimum 2 years (670-1033 days after surgery)
  The Knee Society Score is a self-administered questionnaire. The subject completes questions regarding: Symptoms (3 questions), Patient Satisfaction (5 questions), Patient Expectations (3 questions), Functional Activities (5 questions), Standard Activities (6 questions), Advanced Activities (5 questions), and Discretionary Knee Activities ( 4 questions). The surgeon completes questions regarding objective knee indicators. Likert responses are used, typically with five response options.
Patient Reported Outcome: EuroQol 5D 3L questionnaire (EQ-5D-3L) | Minimum 2 years (670-1033 days after surgery)
  EuroQol 5D 3L questionnaire is a standardized instrument for use as a measure of health outcome that is designed for completion by the subject.
Modified VAS Pain Score: Pain and Satisfaction | Minimum 2 years (670-1033 days after surgery)
  VAS Pain Score is a standardized instrument for use as a measure of pain and satisfaction that is designed for completion by the subject. This modified version has scores that are discrete numbers rather than a continual scale
Type and Frequency of Adverse Events (AEs) for all enrolled subjects | Pre-op (-90 to -1 days before surgery), 6 weeks (1-90 days after surgery), 6 months (91-303 days after surgery), minimum 1 year (304-669 days after surgery), minimum 2 years (670-1033 days after surgery), minimum 5 years (1764-2190 days after surgery)
  All Serious AEs must be reported to Sponsor. All device-related or procedure-related adverse events must be reported to Sponsor.
Survivorship | Minimum 2 years (670-1033 days after surgery)
  Kaplan-Meier survival analysis will be used to calculate the survivorship of all 2 configurations (CR RP, PS RP)
Survivorship | Minimum 5 years (1764-2190 days after surgery)
  Kaplan-Meier survival analysis will be used to calculate the survivorship of all 2 configurations (CR RP, PS RP)
Implant fixation: Radiographic assessment of bone-implant interface performance | 6 weeks (1-90 days after surgery)
  Radiographic success is defined as: absence of progressive radiolucent lines greater than or equal to 2mm in any one zone; absence of lytic lesions in any zone; absence of individual component position change >3degrees in any plane.
Implant fixation: Radiographic assessment of bone-implant interface performance | 6 months (91-303 days after surgery)
  Radiographic success is defined as: absence of progressive radiolucent lines greater than or equal to 2mm in any one zone; absence of lytic lesions in any zone; absence of individual component position change >3degrees in any plane.
Implant fixation: Radiographic assessment of bone-implant interface performance | Minimum 1 year (304-669 days after surgery).
  Radiographic success is defined as: absence of progressive radiolucent lines greater than or equal to 2mm in any one zone; absence of lytic lesions in any zone; absence of individual component position change >3degrees in any plane.
Implant fixation: Radiographic assessment of bone-implant interface performance | Minimum 2 years (670-1033 days after surgery)
  Radiographic success is defined as: absence of progressive radiolucent lines greater than or equal to 2mm in any one zone; absence of lytic lesions in any zone; absence of individual component position change >3degrees in any plane.
Evaluate changes in femoral component and tibial component alignment | Minimum 2 years (670-1033 days after surgery)
  Radiographs will be reviewed by an independent radiographic reviewer (IRR) in order to minimize bias of radiographic outcomes. Data from the IRR radiographic evaluations will be used to evaluate femoral and tibial component alignment over time.

CONTACTS AND LOCATIONS:
Overall Officials: Sukhjeet Kaur, Study Director — Sponsor GmbH
Locations (20):
- United States (10):
  - Colorado Joint Replacement, Denver, Colorado
  - Florida Research Associates, DeLand, Florida
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - New London Hospital, New London, New Hampshire
  - Rothman Institute, Egg Harbor, New Jersey
  - SUNY downstate Medical Center, Brooklyn, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Associated Orthopaedics of Kingsport, Kingsport, Tennessee
  - Texas Tech University Heath Science Center, Lubbock, Texas
  - Hampton Roads Orthopaedics and Sports Medicine, Newport News, Virginia
- Krankenhaus der Barmherzigen Schwestern Ried im Innkreis, Ried im Innkreis, Upper Austria, Austria
- Foothills Medical Centre, University of Calgary, Calgary, Alberta, Canada
- France (2):
  - CHU de la Cavale Blanche, Brest, Cedex
  - Sevice de Chirurgie Orthoedique et Traumatologique, Salouël
- Klinikum Garmisch-Partenkirchen GmbH, Garmisch-Partenkirchen, Germany
- South Infirmary Victoria University Hospital, Cork, Ireland
- Elkerliek Ziekenhuis, Helmond, North Brabant, Netherlands
- University of Otago, Christchurch, New Zealand
- United Kingdom (2):
  - Wrightington Hospital, Wigan, Lancashire
  - Nottingham University Hospitals NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: No